CLINICAL TRIAL: NCT02913183
Title: Efficacy and Safety of Young Health Plasma on Acute Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Xiao-Yi Xiong, Medical Doctor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XinqiaoH-01
Record Dates: First submitted 2016-09-11; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: acute stroke; young health plasma; efficacy; safety
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- young Fresh Frozen Plasma (Experimental): 1. Drug: young plasma will be administered as 2 unit /day over a course of 3 consecutive days after stroke onset.
  2. Drug: young plasma exchange over a course of 3 consecutive days after stroke onset.
  Interventions: Drug: young Fresh Frozen Plasma
- old Fresh Frozen Plasma (Placebo Comparator): 1. Old plasma will be administered as 2 unit /day over a course of 3 consecutive days after stroke onset.
  2. Old plasma exchange over a course of 3 consecutive days after stroke onset.
  3. Patients will receive usual care and drug use in hospital.
  Interventions: Drug: old Fresh Frozen Plasma

INTERVENTIONS:
Drug: young Fresh Frozen Plasma — Blood plasma from healthy male donors aged 18-30 years old.
  Arms: young Fresh Frozen Plasma
Drug: old Fresh Frozen Plasma — Blood plasma from healthy male donors aged 40-55 years old.
  Arms: old Fresh Frozen Plasma

SUMMARY:
Stroke is one of the main severe disease of public health importance. Recent studies showed that old age is one of the most important factors in influencing the outcome of patients with acute stroke, and the young plasma can reverse age-related brain impairments in mice. Therefore, this pilot study aims to investigate whether young plasma is effective in alleviating brain injury and neurologic deficits induced by acute stroke in patients.

DETAILED DESCRIPTION:
This study will enroll 78 stroke patients who have been diagnosed with stroke and meet the inclusion criteria.

After successfully meeting initial screening criteria, investigators will contact the family, explain the study, and send a consent form for their review.

After that, patients will be given 2 unit/day young health plasma (young plasma exchange) over a course of 3 consecutive days, then investigators will make a neurofunctional assessment before and 7 days, 30 days and 90 days after young health plasma treatment. And Magnetic Resonance of the brain before, 7 days, 14 days and 90 days after young health plasma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years
* Clinical presentation of spontaneous intracerebral hemorrhage/ischemic stroke
* CT/MRI/MRA scan compatible with spontaneous intracerebral hemorrhage/ ischemic stroke
* Time to young plasma treatment < 72 h from symptom onset
* Glasgow Coma Score > 6 on initial presentation or improvement to a Glasgow Coma Score > 6 within the time frame for enrollment
* The first-ever primary supratentorial intracerebral basal ganglia hemorrhage 5-30ml
* Signed and dated informed consent is obtained
* TOAST: Large-artery atherosclerosis

Exclusion Criteria:

* Patients who will undergo surgical evacuation of intracerebral hemorrhage/ischemic stroke
* Inability to undergo neuroimaging with Magnetic Resonance
* Glasgow Coma Score < 6
* Significant past history of disability, modified Rankin Scale（mRS）≥1
* Primary intraventricular hemorrhage ICH due to coagulopathy (PT > 15 s or International Normalized Ratio > 1.3, Partial Thromboplastin Time > 36) or trauma
* Thrombocytopenia: platelet count <100 000
* Clinically significant hepatic disease as demonstrated by history, clinical exam (ascites, varices), or laboratory findings (LFTs >2x normal, coagulopathy as described)
* Comorbid conditions likely to complicate therapy including but not limited to the following: a history of New York Heart Association class II, III, or IV Congestive Heart Failure; end-stage acquired immune deficiency syndrome
* Known pregnancy, or positive pregnancy test, or breast feeding
* Malignancy (history of or active)
* Bradyarrhythmia and Atrioventricular Block
* Concomitant use with antineoplastic,immunosuppressive or immune modulating therapies
* Macular Edema
* Life expectancy of less than 90 days due to comorbid conditions
* Occurrences of secondary intracerebral hemorrhage/ischemic stroke
* Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, noncompliance, living in another state or any other cause

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Changes in National Institutes of Health Stroke Scale (NIHSS) | up to 90 days
  describe the clinical improvement at baseline, 7 days, 14 days, 30 days and 90 days
Changes in modified Barthel Index | up to 90 days
  describe the clinical improvement at baseline, 7 days, 14 days, 30 days and 90 days
Changes in modified Rankin Scale | up to 90 days
  describe the clinical improvement at baseline, 7 days, 14 days, 30 days and 90 days
Changes in Glasgow coma scale | up to 90 days
  describe the clinical improvement at baseline, 7 days, 14 days, 30 days and 90 days

SECONDARY OUTCOMES:
Changes in hematoma volume | At baseline, 7 days, 14 days and 30 days after the onset
Change in peripheral edema volume | At baseline, 7 days, 14 days and 30 days after the onset

IPD SHARING:
Plan to Share IPD: Yes
Neurofunctional assessment including NIHSS, modified Barthel Index, modified Rankin Scale,and Glasgow coma scale, hematoma volume,and peripheral edema volume are to be shared.